CLINICAL TRIAL: NCT04922801
Title: OPTIMISING MOLECULAR RADIONUCLIDE THERAPY: The Role of Quantitative SPECT/CT & PET/CT and Radiation Dosimetry (SELFIE)
Brief Title: Optimising Molecular Radionuclide Therapy
Acronym: SELFIE
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS288352
Record Dates: First submitted 2021-05-17; First posted 2021-06-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors; Hyperthyroidism; Thyroid Cancer; Thyroid Carcinoma
Keywords: MRT; Neuroendocrine tumours (NET); 177Lu-DOTATATE; SUV; Quantitative SPECT/CT; Thyroid cancer; I-131; Hyperthyrodism
MeSH Terms: conditions — Neuroendocrine Tumors; Hyperthyroidism; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neuroendocrine Toumours: Patients will undergo 177LU-Dotatate Neoruendocrine Tumours MRT in accordance with existing protocols at GSTTFT. In addition, all MRT patients will be asked to undertake the following non-invasive procedures.
  * Post-treatment gamma camera (Planar Whole Body & SPECT/CT) imaging to estimate disease/ target tissue and whole-body dose for Neuroendocrine and thyroid cancer MRT.
  * Post-treatment gamma camera planar Whole Body imaging for hyperthyroidism MRT.
  * Post-treatment patient-led self-monitoring.
  * Complete a feedback questionnaire relating to the use of self radiation monitoring.
  Interventions: Diagnostic Test: Nuclear Medicine whole-body; Diagnostic Test: SPECT/CT imaging.; Diagnostic Test: PET/CT imaging.; Device: Patient-led radiation monitor (SELFIE); Diagnostic Test: LAB TEST
- Thyroid Cancer: Patients will undergo 131I-Thyroid cancer MRT in accordance with existing protocols at GSTTFT. In addition, all MRT patients will be asked to undertake the following non-invasive procedures.
  * Post-treatment gamma camera (Planar Whole Body & SPECT/CT) imaging to estimate disease/ target tissue and whole-body dose for Neuroendocrine and thyroid cancer MRT.
  * Post-treatment gamma camera planar Whole Body imaging for hyperthyroidism MRT.
  * Post-treatment patient-led self-monitoring.
  * Complete a feedback questionnaire relating to the use of self radiation monitoring.
  Interventions: Diagnostic Test: Nuclear Medicine whole-body; Diagnostic Test: SPECT/CT imaging.; Diagnostic Test: PET/CT imaging.; Device: Patient-led radiation monitor (SELFIE); Diagnostic Test: LAB TEST
- Hyperthyrodism: Patients will undergo 131I-Hyperthyroidism MRT in accordance with existing protocols at GSTTFT. Patients will have one whole-body scan at 24 hr post MRT which will not involve any additional radiation. In addition, all MRT patients will be asked to undertake the following non-invasive procedures.
  * Post-treatment gamma camera (Planar Whole Body & SPECT/CT) imaging to estimate disease/ target tissue and whole-body dose for Neuroendocrine and thyroid cancer MRT.
  * Post-treatment gamma camera planar Whole Body imaging for hyperthyroidism MRT.
  * Post-treatment patient-led self-monitoring.
  * Complete a feedback questionnaire relating to the use of self radiation monitoring.
  Interventions: Diagnostic Test: Nuclear Medicine whole-body; Diagnostic Test: PET/CT imaging.; Device: Patient-led radiation monitor (SELFIE); Diagnostic Test: LAB TEST

INTERVENTIONS:
Diagnostic Test: Nuclear Medicine whole-body — Gamma-Camera Whole-body scan at 24-48 hour post-Molecular Radiotherapy (MRT).
Diagnostic Test: SPECT/CT imaging. — SPECT/CT scan at 24-48 hr post MRT
  Groups: Neuroendocrine Toumours; Thyroid Cancer
Diagnostic Test: PET/CT imaging. — 3-6 months Pre and post-therapy PET/CT imaging
Device: Patient-led radiation monitor (SELFIE) — Following MRT administration, a standard whole body dosimetry measurement will be taken by medical physicist at 1 and 2 meters distance. The patient will begin to take SELFIE readings at the same time under supervision so that their records can be compared with the physicists' results.
  After 28 days, patients will be asked to return the diary sheet and SELFIE monitor by post to GSTTFT in a pre-paid, pre-addressed envelope.
  On completion of the 28 day exercise, patients will be asked to complete and return a feedback questionnaire.
Diagnostic Test: LAB TEST — Biochemistry, haematology and tumour markers blood tests pre, post and during MRT.

SUMMARY:
This project will examine the role of the whole body, PET and SPECT imaging before, during and after radionuclide treatment for 177Lu-Dotatate therapy, whole body and SPECT imaging for 131-I for thyroid cancer therapy, and whole-body imaging for 131I for hyperthyroidism therapy. Whole-body and SPECT images will be linked to personal dosimeter readings to determine whether

* Current radiation protection advice for patients receiving radionuclide treatment is appropriate.
* Radiopharmaceutical retention and/or SUV change in patients undergoing repeated radionuclide treatments.
* Data combined from early (quantitative imaging) and late (whole-body dose rate measurements) could support individual treatment planning for patients undergoing repeated cycles of molecular therapy.

DETAILED DESCRIPTION:
This cohort (retro- & prospective) study will be conducted at Guy's and St Thomas' NHS Foundation Trust (GSTTFT) among patients undergoing MRT. Pre and post-therapy blood tests, treatment administration, whole body and SPECT/PET imaging will be undertaken in strict accordance with existing GSTTFT approved protocols for each type of treatment. With the exception of hyperthyroid patients receiving I-131 therapy, these procedures are all part of the standard of care at GSTT. Hyperthyroid patients will be required to have one whole-body scan at 24hrs post-therapy activity administration in addition to their standard care. This will not result in additional radiation exposure.

The decision to proceed with MRT will have been agreed upon at the relevant multidisciplinary meeting in accordance with current practice guidelines. Pre and post-therapy blood tests, whole body and SPECT/PET imaging will be followed as per current GSTTFT protocols. Patients will be asked to undertake the following:

1. Neuroendocrine tumour and thyroid cancer patients: 1-7 days treatment whole-body gamma camera and SPECT /CT scan. (Part of standard of care post-treatment monitoring at GSTTFT).

   *Hyperthyroid patients: 24-hour post-treatment whole-body gamma camera scan. (Part of this research protocol, will not involve any additional radiation).
2. Record SELFIE reading for 28 days post-therapy using the sheet provided. (Part of this research protocol).
3. Complete feedback questionnaire. (Part of this research protocol). *Benign thyroid disease patients only: Reasonable travel expenses for the cost of an additional hospital visit for post-treatment scans will be reimbursed from the nuclear medicine research fund SPF228. (Maximum reimbursement 50 £)

For the purpose of this study, two dosimetry methods will be used and compared.

1. Whole-body self-monitored retention measurements study (SELFIE study):

   A handheld radiation monitor (ATOMTEX model AT6130, Belarus) will be used to follow the time course of radioactivity clearance in each patient. The measurement device (SELFIE device) will be introduced to patients by a member of the medical physics team. Patients will be shown how to operate and record readings obtained and will also receive illustrated written instructions to build confidence. The devices are user friendly and patients will be asked to record the measurements twice daily using a diary sheet, typically taking about one minute to complete on each occasion. Measurement can begin immediately following administration and will continue for 28 days afterwards.

   Following MRT administration, a standard whole-body dosimetry measurement will be taken by a medical physicist at 1 and 2 meters distance. The patient will begin to take SELFIE readings at the same time under supervision so that their records can be compared with the physicists' results.

   After 28 days, patients will be asked to return the diary sheet and SELFIE monitor by post to GSTTFT in a pre-paid, pre-addressed envelope.

   On completion of the 28-day exercise, patients will be asked to complete and return a feedback questionnaire.

   The paper record of SELFIE readings will be reviewed by investigators from each patient for 28 days post-therapy. All imaging will be performed at GSTTFT by specialist Nuclear Medicine/PET staff.

   All acquired images will be reconstructed and analysed by investigators using HERMES software as described in section 13.3.
2. Imaging response assessment Planar Whole body, SPECT/CT and PET/CT images will be acquired to assess uptake patterns and, in the case of sequential treatments, uptake/retention changes. SPECT/CT, PET/CT and whole-body scans will be performed in accordance with existing protocols at Guy's and St. Thomas' NHS Foundation Trust. This will not result in additional radiation exposure. (Schedule illustrated in 16.1 Appendix).

The SUV of target and non-target tissues will be calculated from quantitative pre and post-therapy PET/CT and post-therapy SPECT/CT images. As a result, early tumour response and toxicity in patients undergoing molecular targeted radionuclide therapy can be studied.

Patient-led dose rate (SELFIE) data and imaging data will be integrated to compare whole-body retention and evaluate sequential dose rate changes after repeated treatments.

The quality of SELFIE data will be assessed against pre-specified standards (completeness of data collection, data deviation). Patient satisfaction will be evaluated from the feedback questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving MRT (177Lu-Peptide for Neuroendocrine Tumours and 131I for Thyroid Cancer and Benign Hyperthyroidism).
* Women of childbearing potential must use a reliable method of contraception and have a documented negative pregnancy test immediately prior to MRT administration in accordance with routine clinical practice.
* Able to comply with treatment plans, scheduled visits, all study whole body, SPECT/CT & PET/CT imaging and follow-up.
* Able to use a personalised dosimetry handheld device and record daily readings for 28 days post MRT.
* Willing and able to give informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Any other considerations that may make the patient unable to tolerate whole body, PET or SPECT scans.
* Inability to use a personalised dosimetry handheld device and record the daily reading for 28 days post MRT.
* Participants who are involved in current research or have recently been involved in any research prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients undergoing molecular radionuclide therapy at GSTTFT using Lutetium-177 peptides for neuroendocrine tumour and I-131 for benign and malignant thyroid disease therapy will be invited to participate.
  The total sample size is estimated as 60 patients divided as 20 for patients receiving 131I for hyperthyroidism, 20 patients for 131I for thyroid cancer and 20 patients for177Lu-DOTATATE for neuroendocrine tumours. This sample should allow sufficient quantitative and dosimetry data to explore the research questions. The range in the number of patients who will be studied is intended to mitigate uncertainty regarding continuing restrictions related to the COVID-19 Coronavirus pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
20 patients with Lu-Dotatate MRT response to therapy outcome as Assessed by response evaluation criteria in solid tumours RECIST (version 1.1) | started from the day of MRT administration at cycle 1 and cycle 4. (Total 4 MRT cycles, each cycle length 8-12 weeks). each participant time frame 1 year.
  * Standardised uptake value (SUV) will be extracted from SPECT/CT image using HERMES software at cycle 1 and cycle 4 of Lu-Dotatate MRT.
  * SUV values will be extracted from PET/CT image Pre and post Lu-Dotatate MRT using HERMES software.
  * The descriptive( mean, max, min, SD) and inferential (Wilcoxon signed-rank test and Spearman correlation) analysis will be applied to calculate the changes in SUV values in SPECT and PET.
  SUV changes will be correlated between SPECT & PET.
Whole-body gamma image time activity curve (TAC) versus patient-led external dose rate (SELFIE) TAC. | SELFIE: 28 days measurements post administration of MRT activity. and Whole-body image:24 hrs post administration of MRT activity.
  The data from both sets will be synthesised from all defined groups in this study to establish if correlation points exist between whole-body imaging and the selfie TAC.
  Nonlinear biexponential curve fitting will be applied using GraphPad statistics software to generate SELFIE slow and fast halflives and TAC.
  Hermes software will be used to generate whole-body gamma image TAC. Spearman correlation will be applied to test correlation.

SECONDARY OUTCOMES:
Patient-led external dose measurement (SELFIE) area under the curve (AUC) change between cycle 1 & 4 MRT | 1 year for Neuroendocrine tumours participants and 1 month for thyroid cancer and hyperthyroidism participants.
  Data will be extracted from SELFIE for 28 days post MRT to generate AUC using biexponential nonlinear curve fitting to evaluate sequential dose rate change after repeated treatment.
MRT patients Acceptance of patient-led monitor (SELFIE) | 28 days post MRT activity administration.
  All MRT groups identified in this study will complete the 5 Likert scale SELFIE Questionnaire (Agreement: Strongly agree, Agree, Neither agree nor disagree, Disagree, Strongly disagree).
  Descriptive analysis and non-parametric tests such as Spearman's correlation or chi-square test for independence for individual Likert-scale questions.
  Questionnaire to be submitted to the research team after 28 days of using SELFIE

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lewington, Professor, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas Hospitals Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: From June 2023 till June 2028.
Access Criteria: IPD will be shared with the lead sponsor King's College London. Name of Sponsor representative: Professor Reza Razavi Address: King's College London Vice President & Vice-Principal (Research) Room 5.31, James Clerk Maxwell Building 57 Waterloo Road London SE1 8WA Telephone: Tel: +44 (0)207 8483224 Email: reza.razavi@kcl.ac.uk
  • Once the project has ended, data that supports published research and/or has long term value will be deposited with the university's research data repository to ensure long term preservation and accessibility. King's is committed to preserving research data for a minimum of 10 years since the last use of the data. Patient's images will be stored at HERMES medical system located in Nuclear Medicine Department at GSTTFT.